CLINICAL TRIAL: NCT07111468
Title: A Multicenter, Randomized, Double-blind, Parallel, Active-controlled, Superiority, Phase III Clinical Trial to Evaluate the Efficacy and Safety of YHP2401 Compared to YHR2402 and YHR2403 for Acute Bronchitis
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of YHP2401 Compared to YHR2402 and YHR2403 for Acute Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YHP2401-301
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YHP2401 (Experimental)
  Interventions: Drug: YHP2401
- YHR2402 (Active Comparator)
  Interventions: Drug: YHR2402
- YHR2403 (Active Comparator)
  Interventions: Drug: YHR2403

INTERVENTIONS:
Drug: YHP2401 — Total 7 days of treatment and The daily dose is tid.(YHP2401 + Placebo of YHR2402 + Placebo of YHR2403)
  Arms: YHP2401
Drug: YHR2402 — Total 7 days of treatment and The daily dose is tid.(Placebo of YHP2401 + YHR2402 + Placebo of YHR2403)
  Arms: YHR2402
Drug: YHR2403 — Total 7 days of treatment and The daily dose is tid.(Placebo of YHP2401 + Placebo of YHR2402 + YHR2403)
  Arms: YHR2403

SUMMARY:
A Multicenter, Randomized, Double-blind, Parallel, Active-controlled, Superiority, Phase III Clinical Trial to Evaluate the Efficacy and Safety of YHP2401 Compared to YHR2402 and YHR2403 for Acute Bronchitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 19 years ≤ age ≤ 80 years
* Patients with acute bronchitis presenting with productive cough symptoms within 48 hours prior to Visit 2 (Baseline)
* BSS total score ≥ 5 at Visit 2, including Cough score ≥ 2, Sputum score ≥ 1
* Patients who voluntarily signed the consent form

Exclusion Criteria:

* Severe lung disease as determined by the investigator
* Clinically significant abnormal findings or signs on chest X-ray suggesting diagnoses other than acute bronchitis
* Active infection requiring systemic antibiotic treatment
* Patients who need to take contraindicated concomitant medications

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Bronchitis Severity Score(BSS) | Day 4

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - Soonchunhyang University Hospital Bucheon, Bucheon-si
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Wonkwang University Hospital, Iksan
  - Kangbuk Samsung Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St.Mary's Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No